CLINICAL TRIAL: NCT01138969
Title: Efficacy of Proton Pump Inhibitor in Prevention of Clopidogrel-related Peptic Ulcer and Gastrointestinal Bleeding
Brief Title: Efficacy of Proton Pump Inhibitor in Prevention of Clopidogrel-related Peptic Ulcer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Chief, Gastroenterology Division, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VGHKS98-CT6-12
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Peptic Ulcer
Keywords: proton pump inhibitor; peptic ulcer; clopidogrel; prevention
MeSH Terms: conditions — Peptic Ulcer | interventions — Esomeprazole; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esomeprazole plus clopidogrel group (Active Comparator): esomeprazole (20 mg qd) plus clopidogrel (75 mg qd) for 6 months
  Interventions: Drug: esomeprazole
- Clopidogrel group (No Intervention): clopidogrel 75 mg qd for 6 months

INTERVENTIONS:
Drug: esomeprazole — esomeprazole 20 mg qd for 6 months
  Other Names: plavix
  Arms: Esomeprazole plus clopidogrel group

SUMMARY:
Proton Pump Inhibitors (PPI) can prevent the recurrence of peptic ulcer in clopidogrel users.

DETAILED DESCRIPTION:
The aim of the prospective, randomized study is to investigate the efficacy of PPI in prevention of ulcer recurrence for clopidogrel users. We plan to enroll 300 clopidogrel users without baseline gastroduodenal ulcer at initial endoscopy. The patients will be randomly assigned to receive either (1) esomeprazole (20 mg qd) plus clopidogrel or (2) clopidogrel treatment alone for 6 months. The ulcer recurrence rate between the treatment groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* We plan to enroll 300 clopidogrel users without baseline gastroduodenal ulcer at initial endoscopy. The patients will be randomly assigned to receive either (1) esomeprazole (20 mg qd) plus clopidogrel or (2) clopidogrel treatment alone for 6 months.

Exclusion Criteria:

* 1.serious disease 2.refuse informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Hung Lai, MD, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Hsu PI, Lai KH, Liu CP. Esomeprazole with clopidogrel reduces peptic ulcer recurrence, compared with clopidogrel alone, in patients with atherosclerosis. Gastroenterology. 2011 Mar;140(3):791-8. doi: 10.1053/j.gastro.2010.11.056. Epub 2010 Dec 7. PMID 21144850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Dates of the recruitment period: From August 2008 to August 2012
  2. Type of location: Kaohsiung Veterans General Hospital
Pre-assignment Details: None were excluded following participant enrollment.
Period: Overall Study
Arm/Group | Esomeprazole Plus Clopidogrel Group | Clopidogrel Group
Started | 83 | 82
Completed | 83 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole Plus Clopidogrel Group | Clopidogrel Group | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 21 | 46
  >=65 years | 58 | 61 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (11.5) | 73.3 (10.7) | 72.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 65 | 59 | 124
Region of Enrollment [Number; unit: participants]
  Taiwan | 83 | 82 | 165

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Peptic Ulcer
Description: Number of participants with recurrent peptic ulcer within 6 months
Time Frame: 6 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Esomeprazole Plus Clopidogrel Group | Clopidogrel Group
Number analyzed (Participants) | 83 | 82
participants | 1 | 9

2. Secondary Outcome: Peptic Ulcer Bleeding
Description: participants with peptic ulcer bleeding within 6 months
Time Frame: 6 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Esomeprazole Plus Clopidogrel Group | Clopidogrel Group
Number analyzed (Participants) | 83 | 82
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Esomeprazole Plus Clopidogrel Group | Clopidogrel Group
Serious Adverse Events (participants affected / at risk) | 2/83 | 2/82
Other Adverse Events (participants affected / at risk) | 1/83 | 1/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole Plus Clopidogrel Group (N=83) | Clopidogrel Group (N=82)
acute myocardial infarct (Cardiac disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole Plus Clopidogrel Group (N=83) | Clopidogrel Group (N=82)
unstable angina (Cardiac disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The patients without symptoms who refused follow-up endoscopy were regarded as having no recurrent ulcers. Because peptic ulcer may be asymptomatic, the cumulative number of recurrent peptic ulcer might be underestimated in both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes